CLINICAL TRIAL: NCT06965712
Title: Use of Point-of-Care Ultrasound (POCUS) to Guide Fluid Management and Reduce Hospital Length of Stay in Patients With Decompensated Heart Failure
Brief Title: Use of Point-of-Care Ultrasound (POCUS) to Reduce Hospital Length of Stay in Patients With Heart Failure ( POCUSHF )
Acronym: POCUSHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-0179
Record Dates: First submitted 2025-04-30; First posted 2025-05-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Decompensated Heart Failure; Hospital Length of Stay
Keywords: Heart Failure; Decompensated Heart Failure; Point-of-Care Ultrasound; POCUS; Hospital Length of Stay; Ultrasound-Guided Therapy; Lung Ultrasound; Inferior Vena Cava Ultrasound; Volume Status Assessment; Readmission Prevention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either a Point-of-Care Ultrasound (POCUS)-guided evaluation group or a standard clinical evaluation group. Participants in each group will remain in their assigned arm throughout the duration of their hospital stay. The study is designed as a parallel assignment model without crossover between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POCUS-Guided Evaluation Group (Experimental): Participants in this group will receive bedside Point-of-Care Ultrasound (POCUS) evaluations of the lungs and inferior vena cava (IVC) twice during hospitalization, once within 24 hours of admission and once prior to discharge. Ultrasound findings will be used to guide fluid management decisions.
  Interventions: Device: Point-of-Care Ultrasound (POCUS)
- Standard Clinical Evaluation Group (No Intervention): Participants in this group will receive standard clinical care without bedside ultrasound guidance. Clinical evaluation and management will be based on physical examination, chest X-rays, laboratory results, and physician judgment.

INTERVENTIONS:
Device: Point-of-Care Ultrasound (POCUS) — Participants assigned to this group will receive Point-of-Care Ultrasound (POCUS) evaluations of the lungs and inferior vena cava (IVC) during their hospital stay. The ultrasound will be performed twice: once within 24 hours of hospital admission and once prior to hospital discharge. The POCUS findings will be used to guide clinical management decisions regarding fluid status and decongestion therapy in patients with decompensated heart failure. The procedure is non-invasive, radiation-free, and performed at the bedside.
  Arms: POCUS-Guided Evaluation Group

SUMMARY:
This study will evaluate whether using bedside ultrasound (also called Point-of-Care Ultrasound or POCUS) can help improve the care of hospitalized patients with decompensated heart failure. Patients will be randomly assigned to two groups: one group will receive ultrasound-guided assessments, and the other group will receive standard clinical evaluations. Researchers will compare the hospital length of stay between the two groups. Ultrasound is a non-invasive, safe, and painless imaging tool. The goal of the study is to find out if ultrasound guidance can lead to shorter hospitalizations and better care for patients with heart failure.

DETAILED DESCRIPTION:
This clinical trial aims to determine whether the use of bedside ultrasound (also called Point-of-Care Ultrasound, or POCUS) can improve the management of patients hospitalized with decompensated heart failure. Traditional methods for assessing heart failure patients rely heavily on physical examination and imaging tests such as chest X-rays, which may not always accurately reflect a patient's volume status. POCUS provides real-time information at the bedside, allowing clinicians to assess lung congestion and venous volume status quickly and non-invasively.

Participants in this study will be randomly assigned to one of two groups. The intervention group will undergo POCUS assessments of the lungs and inferior vena cava (IVC) twice during their hospitalization: once within 24 hours of admission and once before discharge. The control group will receive standard clinical care without ultrasound guidance. All participants' clinical information, including length of hospital stay, treatments administered, and 30-day readmission status, will be collected and analyzed.

The primary objective is to determine whether POCUS-guided management leads to a reduction in hospital length of stay. Secondary objectives include evaluating whether ultrasound guidance affects 30-day readmission rates and diuretic therapy adjustments. The study is expected to enroll approximately 66 patients.

This research may help establish whether POCUS can be incorporated into standard care practices for hospitalized heart failure patients, potentially leading to better outcomes and more efficient use of hospital resources.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years and older.

Hospitalized with a primary diagnosis of decompensated heart failure (left, right, or biventricular).

Evidence of volume overload or congestion based on Framingham criteria, clinical examination, elevated proBNP (>1000 pg/mL), or chest X-ray showing pulmonary edema.

Ability to undergo bedside ultrasound evaluation (POCUS) as clinically feasible.

Able to provide informed consent.

Exclusion Criteria:

Age under 18 years.

Pregnant or breastfeeding women.

Terminal illness with life expectancy < 30 days.

Inability to obtain ultrasound images due to body habitus or other technical reasons.

Enrollment in another interventional clinical trial that could interfere with the outcomes of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Length of Stay (LOS) | From the date of hospital admission to the date of discharge order, assessed up to 30 days.
  Hospital Length of Stay (LOS) will be measured as the number of days from hospital admission to discharge decision. LOS will be compared between the POCUS-guided group and the standard care group.

SECONDARY OUTCOMES:
30-Day Hospital Readmission Rate | Within 30 days after hospital discharge
  The proportion of patients readmitted to any hospital for any cause within 30 days after discharge will be recorded and compared between the POCUS-guided group and the standard care group.

CONTACTS AND LOCATIONS:
Overall Officials: GUILLERMO IZQUIERDO PRETEL, MD, Principal Investigator — Florida International University
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
I am running a single-center investigator-initiated study. I am not creating a formal public repository for the individual patient data.
  At this stage, I am focused on analyzing your results internally (not distributing patient-level data to outside researchers).